CLINICAL TRIAL: NCT00214877
Title: Double-Blind Trial of Methylene Blue for Cognitive Dysfunction in Bipolar Disorder
Brief Title: Methylene Blue for Cognitive Dysfunction in Bipolar Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Stanley Medical Research Institute (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: QE-RS/2002-173; Stanley Foundation # 02T-166
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-03

CONDITIONS: Bipolar Disorder
Keywords: methylene blue for cognitive dysfunction in bipolar disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Methylene Blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Methylene Blue

SUMMARY:
While many bipolar patients treated with mood stabilizing medications experience improvement in their symptoms, some continue to have ongoing difficulties with concentration and memory. The purpose of this study is to look at whether these symptoms can be improved by adding the compound methylene blue to the treatment plan of patients who are already taking lamotrigine.

Methylene blue is an available 'over the counter medication' in Canada. It has been studied in the long-term treatment of mood symptoms in bipolar disorder. Several clinical studies done in bipolar disorder report that methylene blue has had positive effects on both cognition and mood. It is important to do further research in this area as we know that, for patients who continue to have ongoing cognitive difficulties, there is no recognized standard of care for bipolar patients who experience these type of deficits.

DETAILED DESCRIPTION:
This is a double blind cross-over study. There are two dose ranges in this study. A cross over design means that some patients will start at one dose range and others with another. About half way through the study, patients will then be switched over to the other dose range. Patients partially stabilized on lamotrigine will be randomized to either subtherapeutic (16mg) or therapeutic (200mg) dose of methylene blue. This design is necessary because methylene blue stains urine and thus it is not possible to use a traditional placebo. Double-blind means that neither the doctor nor the patient will know which strength of study drug the patient will be on at what point in the study. The study will be conducted in three centres, each recruiting 20 subjects over a two-year period. The duration of the study is 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Men or women between the ages of 18 and 65 who meet both RDC and DSM-IV criteria for bipolar I or bipolar II disorder will be recruited.
* All subjects will be interviewed using SADS interview (40) with added questions as to arrive at DSM-IV diagnoses as well.
* The patients will be treated with lamotrigine as their main mood stabilizer. Patients recruited for the study will show at least partial response to prophylactic treatment with respect to the mood symptoms.
* HAM-D (17 item) scores at study entry will be 15 or lower and Y MRS scores will be less than 15.

Exclusion Criteria:

* Patients not able to give informed consent
* Patients with active substance abuse or dependence or a history of such within the past two years
* Physical illness, mainly liver and kidney disorders and G-6-PD deficiency
* Subjects previously treated with methylene blue
* Pregnant or breast-feeding women
* Subjects who have had ECT within the past two years
* Patients with known brain injury or loss of consciousness of duration greater than ten minutes
* Subjects taking concurrent medications that are known to have cognitive effects (eg. beta blockers)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2003-11; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Young Mania Rating Scale
Hamilton Depression Rating Scale (HAM-D), 17-item version Hamilton Rating Scale for Anxiety (HAM-A).
Clinical Global Impression Scale CGI-BP (41)
Affective Morbidity Index (42)

SECONDARY OUTCOMES:
California Verbal Learning Task and a process dissociation task. Two tasks will focus on selective attention, negative priming and inhibition of return tasks.
A visual backward masking task that has been well studied in patients with BD will be used.
Trails B will be administered as a test of executive function.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Alda, MD FRCPC, Principal Investigator — Dalhousie University
Locations (2):
- Canada (2):
  - CDHA- QE II Health Sciences Centre, Halifax, Nova Scotia
  - St. Joseph's Healthcare, Hamilton, Ontario

REFERENCES:
- [Derived] Alda M, McKinnon M, Blagdon R, Garnham J, MacLellan S, O'Donovan C, Hajek T, Nair C, Dursun S, MacQueen G. Methylene blue treatment for residual symptoms of bipolar disorder: randomised crossover study. Br J Psychiatry. 2017 Jan;210(1):54-60. doi: 10.1192/bjp.bp.115.173930. Epub 2016 Jun 9. PMID 27284082